CLINICAL TRIAL: NCT01404377
Title: Double Blind Randomized Trial of Wound Infiltration With Ropivacaine After Breast Cancer Surgery
Brief Title: Wound Infiltration and Breast Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tenon Hospital, Paris (Other)
Responsible Party: F Bonnet, association pour la recherche en anesthésie réanimation hôpital Tenon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TenonH; bordereau 52 rang 5 N°338 (Other: Direction Regionale des affaires sanitaires et sociales)
Record Dates: First submitted 2011-04-11; First posted 2011-07-28 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
Keywords: breast surgery : postoperative pain; ropivacaine
MeSH Terms: conditions — Breast Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine (Active Comparator): treated group (ropivacaine infiltration)
  Interventions: Procedure: infiltration with ropivacaine solution
- placebo (Placebo Comparator): placebo group : infiltration with saline solution
  Interventions: Procedure: infiltration with ropivacaine solution

INTERVENTIONS:
Procedure: infiltration with ropivacaine solution — Patients are allocated randomly into two arms on the morning of surgery, using random numbers and sealed envelopes. In the treated group infiltration is performed with a ropivacaine 7.5 mg.ml-1 solution and in the control group with an isotonic saline solution. In the two groups patients are operated under and nitrous oxide for maintenance. Dexamethasone 4 mg was given intravenously after anaesthetic induction for prevention of postoperative nausea and vomiting. Twenty milliliters of the allocated solution were used at the end of the surgical procedure to infiltrate the subcutaneous and deep layers at the level of the breast and axilla surgical incision.
  Other Names: naropeine

SUMMARY:
Prospective double blind randomized evaluation of the effect of surgical wound infiltration with ropivacaine versus placebo in patients scheduled for breast surgery with axillary lymph node dissection

DETAILED DESCRIPTION:
This is a prospective, double-blind, randomized, single centre study Adult ASA I - II patients, scheduled for unilateral mastectomy or tumorectomy associated with axillary lymph node dissection are included in the study. Patients receiving opioid or any other analgesic treatment for chronic pain before surgery, patients with known allergy to local anaesthetics, and patients with acquired or genetic haemostatic abnormality are excluded.

Patients are allocated randomly into two groups on the morning of surgery, using random numbers and sealed envelopes. general anaesthesia using propofol and sufentanil for induction, and sevoflurane In the treated group infiltration is performed with a ropivacaine 7.5 mg.ml-1 solution and in the control group with an isotonic saline solution. In the two groups patients are operated under general anesthesia with propofol, sufentanil, sevoflurane and nitrous oxide for maintenance. Twenty milliliters of the allocated solution are used at the end of the surgical procedure to infiltrate the subcutaneous and deep layers at the level of the breast and axilla surgical incision. Postoperatively, 8 tablets of paracetamol 500 mg were let at patient' disposal every 24 hours for 3 days. If pain control is not adequate patients receive 5 mg of subcutaneous morphine as a rescue.

Pain intensity is measured on a visual analogue scale graded from 0 to 100. Measurements are performed at rest and on operated arm abduction, at 2, 4, 6, 12, 24, 48, and 72 hour after the end of surgery. The value of maximum abduction angle is noted.

To evaluate quality of life patients are asked to score on a 4 points scale graded from 0 (the worst) to 3 (the best) the following items: sleep - fatigue - global activity - relationship with relatives - state of mood. A global score is attributed to each patient as the sum of categorical scores. Evaluation is performed at 24, 48 and 72 hour after the end of surgery.

Patients are evaluated at two month for residual pain at rest and on movement using a visual analogue scale and for quality of life as previously defined.

ELIGIBILITY:
Inclusion Criteria:

* Adult ASA I - II patients, scheduled for unilateral mastectomy or tumorectomy associated with axillary lymph node dissection

Exclusion Criteria:

* Patients receiving opioid or any other analgesic treatment for chronic pain before surgery, patients with known allergy to local anaesthetics, and patients with acquired or genetic haemostatic abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
30% decrease in VAS score on mobilization on the day of surgery | patients will be followed during all the duration of hospital stay and 2 months after surgery
  Pain intensity was measured on a VAS graded from 0 to 100, on operated arm at maximum abduction, at 2, 4, 6, 12, 24, 48, and 72 hour after the end of surgery.

SECONDARY OUTCOMES:
decrease in pain score at rest | duration of hospitalisation and 2 month after surgery
  Pain intensity was measured on a VAS graded from 0 to 100, at rest at 2, 4, 6, 12, 24, 48, and 72 hour after the end of surgery.
decrease in analgesic rescue consumption | during hospital stay
  patients received non opioid analgesic (paracetamol) on demand postoperatively
improvement in quality of life scoring | during hospital stay
  Quality of life was scored on a 4 points scale graded from 0 (the worst) to 3 (the best) for the following items: sleep - fatigue - global activity - relationship with relatives - state of mood. Evaluation was performed at 24, 48 and 72 hour after the end of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Francis Bonnet, MD, Principal Investigator — Tenon Hospital
Locations (1):
- Hopital Tenon, Paris, France

REFERENCES:
- [Derived] Vigneau A, Salengro A, Berger J, Rouzier R, Barranger E, Marret E, Bonnet F. A double blind randomized trial of wound infiltration with ropivacaine after breast cancer surgery with axillary nodes dissection. BMC Anesthesiol. 2011 Nov 24;11:23. doi: 10.1186/1471-2253-11-23. PMID 22114900